CLINICAL TRIAL: NCT01319695
Title: Corifollitropin Alfa Versus Recombinant Follicle Stimulating Hormone (FSH) in Ovarian Stimulation of Women Undergoing in Vitro Fertilisation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Siristatidis Charalampos, MD, PhD, Assistant Professor, Director of the ARU, National and Kapodistrian University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1234560
Record Dates: First submitted 2011-03-08; First posted 2011-03-22 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2016-04

CONDITIONS: Infertility
Keywords: corifollitropin alfa; FSH ovarian stimulation; IVF
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- corifollitropin alfa (Experimental)
  Interventions: Drug: corifollitropin alfa
- recombinant follicle stimulating hormone (FSH) (Active Comparator): 150-300 IU of FSH for ovarian stimulation in women undergoing IVF
  Interventions: Drug: recombinant follicle stimulating hormone (FSH)

INTERVENTIONS:
Drug: corifollitropin alfa — 100 microg for a group of women weighing <or=60 kg and 150 microg for a group of women weighing >60 kg
  Arms: corifollitropin alfa
Drug: recombinant follicle stimulating hormone (FSH) — 150-300 IU of the drug daily from day 2 of the menstrual cycle until more than 2 follicles are >18mm
  Arms: recombinant follicle stimulating hormone (FSH)

SUMMARY:
The use of corifollitropin alfa is superior in terms of pregnancy outcome parameters as compared to recombinant follicle stimulating hormone (FSH) during ovarian stimulation protocols in women undergoing in vitro fertilisation.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-36 years old with a body weight of more than 60 kg up to 90 kg
* BMI of 18-32 kg/m2
* Menstrual cycle length of 23-35 days
* An indication for controlled ovarian stimulation for IVF or ICSI

Exclusion Criteria:

* history of an endocrine abnormality
* abnormal outcome of blood biochemistry or hematology
* abnormal cervical smear
* chronic disease
* uterine pathology that interfering with the COS treatment (e.g. fibroids ≥ 5 cm)

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2011-01; Primary Completion 2016-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
no of oocytes (>2 between groups) | at egg recovery, through study completion, an average of 2 years

SECONDARY OUTCOMES:
Clinical pregnancy rate cancellation rate miscarriage rate ectopic pregnancy rate | 3 weeks after embryo transfer
  The presence of fetal heart at transvaginal ultrasound at 6+2 gestational weeks
Ongoing pregnancy rate | 12 weeks after embryo transfer
  The presence of fetal heart at ultrasound after 12 gestational weeks
miscarriage rate | through study completion, an average of 2 years
live birth rate | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - 3rd Department of Obstetrics and Gynecology, Assisted Reproduction Unit, Athens, Chaidari
  - Attikon University Hospital, Athens, Chaidari

IPD SHARING:
Plan to Share IPD: Undecided
We will be happy to share the data

REFERENCES:
- [Result] Siristatidis C, Dafopoulos K, Christoforidis N, Anifandis G, Pergialiotis V, Papantoniou N. Corifollitropin alfa compared with follitropin beta in GnRH-antagonist ovarian stimulation protocols in an unselected population undergoing IVF/ICSI. Gynecol Endocrinol. 2017 Dec;33(12):968-971. doi: 10.1080/09513590.2017.1323203. Epub 2017 May 16. PMID 28508691